CLINICAL TRIAL: NCT04733560
Title: Preoperative Analgesia by Infiltration of the Pudendal Nerve Prior to Sacrospinous Ligament Suspension: The PAIN-S Trial
Brief Title: Preoperative Analgesia by Infiltration of the Pudendal Nerve Prior to Sacrospinous Ligament Suspension
Acronym: PAINS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fraser Health (Other)
Responsible Party: Principal Investigator, Sophia Badowski, Principal Investigator, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FHREB2020-143
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Care Provider
Masking Description: Patients are surgeons are blinded to the contents of the injections (either local anesthetic or saline). Allocations will be revealed after all data is collected at the time of data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pudendal nerve block (Experimental): 25 women will receive pudendal nerve blocks of 0.25% Bupivicaine 10ml administered vaginally prior to making any surgical incisions.
  Interventions: Procedure: Pudendal nerve block; Drug: Bupivacaine Injectable Product
- Placebo (Sham Comparator): 25 women will receive sham pudendal nerve blocks using normal saline. These will also be administed vaginally prior to making any surgical incisions.
  Interventions: Procedure: Sham Pudendal nerve block

INTERVENTIONS:
Procedure: Pudendal nerve block — Vaginally administered pudendal nerve block of 10ml 0.25% Bupivacaine prior to making any surgical incisions.
  Arms: Pudendal nerve block
Procedure: Sham Pudendal nerve block — Vaginally administered pudendal nerve block of 10ml Normal Saline prior to making any surgical incisions.
  Arms: Placebo
Drug: Bupivacaine Injectable Product — Used for pudendal nerve block in the intervention arm
  Arms: Pudendal nerve block

SUMMARY:
Pelvic organ prolapse is a common problem. It affects about half of women and causes uncomfortable bulge sensations (similar to sitting on a ball), urine and stool problems, difficulty with sexual activity and embarrassment. Almost one of every five women undergoes surgery to treat prolapse.Typically, vaginal surgery is done while patients are asleep and local anesthetic- freezing medication- is injected where incisions are made to minimize the pain from surgery when waking up.

Pudendal blocks are nerve blocks where local anesthetic is used to freeze a nerve that supplies sensation to the vulva and vaginal area. It is traditionally used to help with pain for women giving birth, but hasn't been studied well in women undergoing vaginal surgery for prolapse.

The investigators believe that by using a small amount of freezing to provide a pudendal block at the time of surgery, on top of the freezing typically provided, that there will be minimized pain after surgery and improve the recovery process. Based on previous studies using pudendal blocks for different vulvar and vaginal procedures, the investigators believe this to be a safe and potentially beneficial practice.

The investigators are planning to conduct a randomized controlled trial of 50 women. 25 will receive pudendal nerve blocks at the time of surgery, and 25 will receive placebo injections.The investigators will monitor their pain scores, satisfaction, use of pain medications and return to activities in order to determine if our intervention has caused a significant improvement in recovery.

DETAILED DESCRIPTION:
Study Procedures:

Randomization and Blinding:

Women will be randomized to receive either Bupivacaine 0.25% or Normal Saline pudendal injections based on the label within a sealed envelope randomly selected on the day of their surgery. Fifty labels will be created with twenty-five labels each of "Bupivacaine 20ml" or "Normal Saline 20ml" written on them. These will be placed in blank, identical envelopes and sealed and shuffled prior to the start of the study. Upon selection, the sealed envelope will be given to the circulating nurse who will draw up the selected solution and label it "pudendal block". The circulating nurse will be directed to not disclose the contents of the envelope or syringe to the participant or to any other member of the team. They will then re-seal the envelope with tape, place a patient label on it and return it to the surgical team post procedure to be returned to a locked file cabinet within the surgical office at the end of the day, to be kept securely with medical records. Group allocation envelopes will be opened after the collection of all outcome data is complete to allow for data analysis. In order to avoid local anesthetic toxicity, any calculations for other anesthetic agents utilized for the surgical procedure or anesthetic will assume that 20 ml of 0.25% Bupivacaine was administered. In the event that an emergent adverse complication is identified which may be attributable to the administered agent, the treatment allocation can be unblinded if this is deemed clinically necessary by the investigator or other treating physician. In the event this is required, the patient will be withdrawn from the study and excluded from the final analysis, but such case(s) will be described in the final study results.

The circulating nurse already draws up local anesthetic and normal saline as a routine part of this procedure for use in other ways, and so the investigators do not anticipate that their participation in this study will be a large burden of work. The investigators estimate that it will add no more than 2 minutes to their preparation time for the surgery.

Pudendal Block administration:

The Pudendal block will be administered by the Surgeon or Surgical Fellow after the administration of anesthetic and preparation for surgery but before the first surgical incision. It will be administered with standard transvaginal technique.

Standardization of the Anesthesia, Pre-op and postoperative pain management:

Pre-operative, postoperative and intra-operative care will be standardized according to guidelines that meet criteria for current standard of care as outlined in the appendix. These pages will be printed on the chart to identify the patient as a participant in the study and also to remind the surgical and anesthetic team of the guidelines of the study.

Standardization of postoperative pain management after discharge:

All patients will receive the same instructions for management of postoperative pain. They will receive instructions to use acetaminophen (Tylenol) regularly as well as Ibuprofen (Advil) regularly as long as they have no contraindications or allergies to these medications. They will be given a standardized prescription for tramadol to use in addition to these medications for management of breakthrough pain.

Study and Follow up Visits:

The patient will have no additional visits attributed to their participation in this study. Instead they will receive electronic (email or text) surveys and telephone reminders over a period of 2 weeks after their operation. The first survey will take less than 1 minute to complete, the second will take less than 5 minutes to complete, and the final survey less than 10 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Diagnosed with prolapse and planning to undergo vaginal day surgery as treatment.
* Must be undergoing a sacrospinous ligament fixation as part of their procedure. Those undergoing a concurrent anterior and/or posterior vaginal repair, or mid-urethral sling will also be included.
* Able to read and write in English
* Able to complete email surveys for the first 2 weeks after surgery

Exclusion Criteria:

* Those with an allergy to local anesthetic (freezing injections)
* Those who prefer to have surgery under spinal anesthesia
* Those with planned concurrent vulvar, laparoscopic or abdominal surgery, or any planned concurrent vaginal surgery other than those in the inclusion criteria.
* Those with a pre-existing chronic pain disorder requiring the regular use of opioid analgesics (more than twice weekly)
* Those with a history of substance abuse
* Those with a history of bleeding disorder
* Those who would prefer not to participate in the study,
* If unable to receive emails in order to fill out the surveys.
* Inability to provide informed consent
* Currently enrolled in any other research study involving drugs or devices

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Post-operative Pain Score | measured at post-operative day 0
  measured on a Visual Analog scale (1-10)
Post-operative Pain Score | measured at post-operative day 1
  measured on a Visual Analog scale (1-10)
Post-operative Pain Score | measured at post-operative day 14
  measured on a Visual Analog scale (1-10)

SECONDARY OUTCOMES:
Readiness for discharge | measured at post-operative day 0 prior to discharge
  measured on a 5 point Likert scale
Patient satisfaction | measured at postoperative day 0
  measured on a 5 point Likert scale
Patient satisfaction | measured at postoperative day 1
  measured on a 5 point Likert scale
Patient satisfaction | measured at postoperative day 14
  measured on a 5 point Likert scale
Functional Recovery Index | measured at postoperative day 1
  Validated tool by Wong et al. Involving measures of return to activities of daily living
Functional Recovery Index | measured at postoperative day 14
  Validated tool by Wong et al. Involving measures of return to activities of daily living
Post-operative Analgesic use | measured at postoperative day 14
  pill count

CONTACTS AND LOCATIONS:
Locations (1):
- City Centre Obstetrics and Gynecology, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided